CLINICAL TRIAL: NCT00488774
Title: A Phase 2/3 Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of Golimumab Induction Therapy, Administered Intravenously, in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: An Efficacy and Safety Study of Golimumab in Participants With Ulcerative Colitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Protocol was cancelled by company based on overall efficacy, no safety concern
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014188; C0524T16 (Other: Janssen Research & Development, LLC); 2006-003397-94 (Other: Janssen Research & Development, LLC); NCT01842152 (obsolete NCT alias)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-04

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, ulcerative; Golimumab; CNTO 148
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Matching placebo for golimumab, intravenous (IV) (through a vein in the arm) infusion administered at Week 0
  Interventions: Other: Placebo
- Golimumab 1 milligram (mg) per kilogram (kg) (Experimental): Golimumab 1 mg per kg intravenous (IV) infusion administered at Week 0.
  Interventions: Drug: Golimumab 1 mg per kg
- Golimumab 2 mg per kg (Experimental): Golimumab 2 mg per kg intravenous (IV) infusion administered at Week 0.
  Interventions: Drug: Golimumab 2 mg per kg
- Golimumab 4 mg per kg (Experimental): Golimumab 4 mg per kg, intravenous (IV) infusion administered at Week 0.
  Interventions: Drug: Golimumab 4 mg per kg

INTERVENTIONS:
Other: Placebo — Matching placebo for golimumab, intravenous infusion administered at Week 0
  Arms: Placebo
Drug: Golimumab 1 mg per kg — Golimumab 1 mg per kg intravenous (IV) infusion administered at Week 0
  Other Names: CNTO 148
  Arms: Golimumab 1 milligram (mg) per kilogram (kg)
Drug: Golimumab 2 mg per kg — Golimumab 2 mg per kg intravenous (IV) infusion administered at Week 0
  Other Names: CNTO 148
  Arms: Golimumab 2 mg per kg
Drug: Golimumab 4 mg per kg — Golimumab 4 mg per kg intravenous (IV) infusion at Week 0
  Arms: Golimumab 4 mg per kg

SUMMARY:
The purpose of this study is to assess the effects (good and bad) of golimumab (CNTO 148) therapy in participants with active ulcerative colitis (UC) (sores in the colon).

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), double-blind (neither the Physician nor the participant know about the study medication), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), parallel-group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions [treatments]) study to evaluate an appropriate intravenous (through a vein in the arm) golimumab induction dose and to demonstrate the safety and efficacy of intravenous induction dosing with golimumab in participants with moderately to severely active UC. At Week 6, participants will be asked to participate in an additional 1-year maintenance study. Participants not entering the 1-year golimumab maintenance study will be evaluated for safety at Week 16. The duration of study will be 6 weeks for participants who enter the 1-year golimumab maintenance study and 16 weeks for participant who do not enter the 1-year golimumab maintenance study.There are 2 parts in this study. Part 1 is Phase 2 "dose-ranging" portion of study. Participants enrolled in Part 1, will receive a single intravenous infusion of either matching placebo for golimumab or 1 milligram (mg) per kilogram(kg), 2 mg per kg or 4 mg per kg of golimumab. Part 2 of the study is called "dose-confirming" and newly enrolled participants will receive same doses studied in Part 1, until the doses for Part 2 are selected and Phase 3 begins. At the time that the final doses are selected, all newly enrolled participants will receive 1 of the selected doses or matching placebo; this is the start of the Phase 3 portion of the study. Participants will primarily be assessed using Mayo Score (it is a score developed for measuring disease activity). Participants' safety and quality of life will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with moderately to severely active ulcerative colitis (UC) defined by a Mayo score of 6 to 12 inclusive at Baseline (Week 0), including an endoscopic (examination of an internal part of the body with a lighted tube; looking at a part of the body with a lighted tube) subscore of greater than or equal to 2
* Participants must have biopsy results (collected at the screening endoscopy (procedure or obtained within the last year) consistent with the diagnosis of UC
* Participants either currently receiving treatment with, or have a history of failure to respond to, or tolerate, at least 1 of the following therapies: oral 5-aminosalicylate (5-ASAs), oral corticosteroids, 6-mercaptopurine (6-MP) and azathioprine (AZA)
* Participants with current dependency or with a history of corticosteroid dependency (i.e. an inability to successfully taper corticosteroids without a return of the symptoms of UC) - Not have a diagnosis of active TB

Exclusion Criteria:

* Participants with previous exposure to biologic anti-tumor necrosis factor (TNF) agents
* Participants with severe extensive UC that is likely to require a colectomy (surgery to remove part or all of the colon) within 12 weeks of study entry
* Participants having UC limited to the rectum only or to less than 20 centimeter (cm) of the colon
* Presence of a stoma (an artificial permanent opening especially in the abdominal wall made in surgical procedures) or presence of a fistula
* Participants with a history of extensive colonic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (108):
- United States (36):
  - Orange, California
  - Roseville, California
  - Littleton, Colorado
  - Bristol, Connecticut
  - Tampa, Florida
  - Fort Dodge, Iowa
  - Topeka, Kansas
  - Louisville, Kentucky
  - Laurel, Maryland
  - Dearborn, Michigan
  - Troy, Michigan
  - Mexico, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Great Neck, New York
  - Huntington, New York
  - New York, New York
  - Charlotte, North Carolina
  - Kinston, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Galveston, Texas
  - Burlington, Vermont
  - Christiansburg, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (3):
  - Adelaide
  - Brisbane
  - Malvern
- Innsbruck, Austria
- Belgium (2):
  - Bonheiden
  - Leuven
- Bulgaria (2):
  - Rousse
  - Varna
- Canada (8):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- France (3):
  - Clichy
  - Lille
  - Nice
- Germany (4):
  - Hamburg, Hamburg
  - Berlin, State of Berlin
  - Herne
  - Magdeburg
- Hungary (8):
  - Békéscsaba
  - Budapest
  - Gyõr
  - Gyulai Ut 18
  - Miskolc
  - Pécs
  - Székesfehérvár
  - Szombathely
- India (5):
  - Hyderabad Andh Prad
  - Jaipur
  - Lucknow
  - Ludhiana
  - Pune
- Israel (5):
  - Afula
  - Hedera
  - Jerusalem
  - Kfar Saba
  - Tel Aviv
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius LT
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Leiden
  - Rotterdam
- New Zealand (2):
  - Auckland
  - Hastings
- Poland (6):
  - Bialystok
  - Częstochowa
  - Krakow
  - Lodz
  - Skierniewice
  - Sopot
- Romania (2):
  - Bucharest
  - Timișoara
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Belgrade, Serbia
- Slovakia (3):
  - Bratislava
  - Nitra
  - Prešov
- Gothenburg, Sweden
- Ukraine (4):
  - Donetsk
  - Ivano
  - Kiev
  - Vynnytsya

REFERENCES:
- [Derived] Adedokun OJ, Xu Z, Liao S, Strauss R, Reinisch W, Feagan BG, Sandborn WJ. Population Pharmacokinetics and Exposure-Response Modeling of Golimumab in Adults With Moderately to Severely Active Ulcerative Colitis. Clin Ther. 2020 Jan;42(1):157-174.e4. doi: 10.1016/j.clinthera.2019.11.010. Epub 2020 Jan 22. PMID 31982148
- [Derived] Rutgeerts P, Feagan BG, Marano CW, Padgett L, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Zhang H, Colombel JF, Reinisch W, Gibson PR, Sandborn WJ; PURSUIT-IV study group. Randomised clinical trial: a placebo-controlled study of intravenous golimumab induction therapy for ulcerative colitis. Aliment Pharmacol Ther. 2015 Sep;42(5):504-14. doi: 10.1111/apt.13291. Epub 2015 Jun 29. PMID 26119226

RESULTS

PARTICIPANT FLOW:
Groups:
- Golimumab 1 Milligram (mg) Per Kilogram (kg): Golimumab 1 mg per kg intavenous infusion was administered at Week 0.
- Golimumab 2 mg Per kg: Golimumab 2 mg per kg intravenous infusion was administered at Week 0.
- Golimumab 4 mg Per kg: Golimumab 4 mg per kg intavenous infusion was administered at Week 0.
Period: Overall Study
Arm/Group | Placebo | Golimumab 1 Milligram (mg) Per Kilogram (kg) | Golimumab 2 mg Per kg | Golimumab 4 mg Per kg
Started | 77 | 62 | 75 | 77
Completed | 69 | 57 | 70 | 74
Not Completed | 8 | 5 | 5 | 3
Not completed — Withdrawal of consent | 2 | 2 | 2 | 0
Not completed — Other | 6 | 3 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Golimumab 1 mg Per kg: Golimumab 1 mg per kg intavenous infusion was administered at Week 0.
- Total: Total of all reporting groups
Arm/Group | Placebo | Golimumab 1 mg Per kg | Golimumab 2 mg Per kg | Golimumab 4 mg Per kg | Total
Number analyzed (Participants) | 77 | 62 | 75 | 77 | 291
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (12.58) | 40.7 (15.51) | 42.3 (13.14) | 39.9 (14.07) | 41 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 39 | 27 | 117
  Male | 47 | 41 | 36 | 50 | 174

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: Clinical response is defined as decrease from baseline in Mayo score by greater than or equal to 30 percent and greater than or equal to 3, with either a decrease from baseline in rectal bleeding sub-score of greater than or equal to 1 or a rectal bleeding sub-score of 0 or 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and a physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12.
Time Frame: Week 6
Population: The efficay analysis population included all the participants who were randomly assigned to receive study medication. Here 'N' signifies participants who were evaluated for this outcome measure.
Measure: Number; unit: Participants
Groups:
- Golimumab 1 mg Per kg: Golimumab 1 mg per kg intravenous infusion was administered at Week 0.
- Golimumab 4 mg Per kg: Golimumab 4 mg per kg intravenous infusion was administered at Week 0.
Arm/Group | Placebo | Golimumab 1 mg Per kg | Golimumab 2 mg Per kg | Golimumab 4 mg Per kg
Number analyzed (Participants) | 73 | 61 | 75 | 77
Participants | 22 | 22 | 33 | 32
Statistical Analysis 1: Comparison: Placebo vs Golimumab 1 mg Per kg; Test type: Superiority or Other; p = 0.467, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Golimumab 2 mg Per kg; Test type: Superiority or Other; p = 0.081, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Golimumab 4 mg Per kg; Test type: Superiority or Other; p = 0.145, Chi-squared

2. Secondary Outcome: Number of Participants With Clinical Remission
Description: Clinical remission is defined as a Mayo score of less than or equal to 2, with no individual sub-score greater than 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and a physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Golimumab 1 mg Per kg | Golimumab 2 mg Per kg | Golimumab 4 mg Per kg
Number analyzed (Participants) | 73 | 61 | 75 | 77
Participants | 8 | 6 | 12 | 10
Statistical Analysis 1: Comparison: Placebo vs Golimumab 1 mg Per kg; Test type: Superiority or Other; p = 0.832, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Golimumab 2 mg Per kg; Test type: Superiority or Other; p = 0.370, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Golimumab 4 mg Per kg; Test type: Superiority or Other; p = 0.702, Chi-squared

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Arm/Group | Placebo | Golimumab 1 mg Per kg | Golimumab 2 mg Per kg | Golimumab 4 mg Per kg
Serious Adverse Events (participants affected / at risk) | 3/77 | 2/63 | 3/74 | 3/76
Other Adverse Events (participants affected / at risk) | 15/77 | 13/63 | 15/74 | 9/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Golimumab 1 mg Per kg (N=63) | Golimumab 2 mg Per kg (N=74) | Golimumab 4 mg Per kg (N=76)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Golimumab 1 mg Per kg (N=63) | Golimumab 2 mg Per kg (N=74) | Golimumab 4 mg Per kg (N=76)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Fatigue (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1
Haematocrit decreased (Investigations) | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Data collection was not considered complete for primary outcome measure because study was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Twelve months after study ends, Sponsor will be provided with a copy of materials at least 45 days prior to submission, with details of proposed date, journal or conference name of publication & it will have 30 days post receipt to send written request that publication be delayed on the basis it exposes intellectual property that requires propriety protection but it will be only for 60 days after which Investigator will be free to publish. The participation of Sponsor will be acknowledged.